CLINICAL TRIAL: NCT05714046
Title: Effects of a Telerehabilitation Program Based on Yoga Training on Core Stabilization and Physical Fitness in Tennis Players
Brief Title: Telerehabilitation Program Based on Yoga Training in Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-847
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Sports Physical Therapy
Keywords: Tennis; Yoga; Core stabilization; Physical fitness; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: Controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): In addition to routine tennis training yoga exercise training was applied to the yoga group 2 days a week for 8 weeks with the telerehabilitation method.
  Interventions: Behavioral: Yoga training
- Control Group (Experimental): Routine Tennis training and information training was given to Control group.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Control — An informative presentation
  Arms: Control Group
Behavioral: Yoga training — Yoga exercise training
  Arms: Yoga Group

SUMMARY:
Although there are frequent studies on core strength in tennis players in the literature, studies on exercise applications targeting the development of physical fitness parameters are limited. In this context, it was aimed to investigate the effect of telerehabilitation method and yoga exercise practice on core stabilization and physical fitness.

DETAILED DESCRIPTION:
Core training is mostly used to improve balance, strength, functional alignment and flexibility. Core training can be a good option to improve physical fitness parameters. It has been observed that core stability training improves core function and trunk control, and positively affects functional and trunk flexibility.

It has been shown that the flexibility of people who practice yoga regularly increases, their posture improves, the mobility of the joints increases, the muscles become stronger, the stability of the ligaments increase, the kinetic chain load transfer is more effective, the breath control is formed, and the person feels more free and dynamic. The target areas of poses such as downward facing dog, plank, boat, shoulder pose, bakasana, which are among the yoga poses, are the core region of the body and are movements that develop core muscles with core activation. Many of the yoga poses require body physical fitness parameters to maintain the pose.

In order for individuals to continue their rehabilitation processes in their own environment and to participate in their training, the telerehabilitation system was frequently used, and according to the results of the study, the effectiveness of the practices performed with telerehabilitation was found to be at a high level.

In this study, it was aimed to investigate the effect of telerehabilitation method and yoga exercise practice on core stabilization and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* Have been playing tennis for at least one year
* Healthy individuals without chronic disease
* No acute injury
* Training at least 4 hours a week
* Using computer and internet

Exclusion Criteria:

* Surgery within the last 6 months
* Having a neurological disease
* Having musculoskeletal diseases
* Use of stimulants
* Use of drugs that will affect psychological or balance
* Inability to use a computer
* Not having internet access

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
Sport-specific core muscle strength and stability test. | 0-8 weeks
  This test, which aims to measure the core strength and endurance of athletes, consists of 8 stages. The time to stay fixed in 8 different positions was calculated while the athlete was in the plank position on his elbows.

SECONDARY OUTCOMES:
Back scratch test | 0-8 weeks
  The athlete was asked to bring his fingers closer so that the palm of one hand was facing the back of the other hand. The distance between the middle fingertips of both hands was measured.
Sit-reach test | 0-8 weeks
  The athlete was positioned in a long sitting position on the floor with bare feet and comfortable clothes, with the ankle in neutral position. The athlete was asked to bend forward in two from the groin, to reach as far as he could go without bending his knees, and to stay at that last point for two seconds. Measurements were performed in duplicate and the best score was recorded in centimeters.
Flamingo test | 0-8 weeks
  The athlete was asked to stand on the 15 cm long and 4 cm wide wooden plate with his dominant foot, bend the other foot from the knee, pull it towards his hip, hold his foot with the same hand and remain in balance for 1 minute. Whenever the balance was disturbed, the timer was stopped, when the balance was restored, the timer was started again and the number of falls per minute was noted.
Y balance test-lower quadrant | 0-8 weeks
  The individual was asked to stand on one foot at the midpoint of the test setup consisting of Y-shaped tapes, and to touch the other foot with the tip of the toe in the anterior, posteromedial and posterolateral directions. The test was repeated 3 times in all directions and the average was taken.
Upper extremity closed kinetic chain stability test | 0-8 weeks
  The athlete took a push-up position between two lines marked on the floor at a distance of 91.4 cm, feet shoulder-width apart, spine and legs lined up in a straight line. The athlete touched the two end points of the line with his hands alternately and quickly for 15 seconds. 3 repetitions were made and the average touch was calculated.
Short form-36 | 0-8 weeks
  The questionnaire consists of 36 items questioning the quality of life in eight sub-dimensions. Subscales evaluate health between 0-100 and the higher the score, the better the quality of life.
Body awareness questionnaire | 0-8 weeks
  It consists of four subgroups and a total of 18 statements aimed at determining the normal or abnormal sensitivity level of body composition. The participant was asked to score a number between 1 and 7 for each statement. Higher score indicated better body responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)